CLINICAL TRIAL: NCT01160757
Title: A Study to Determine the Safety and Efficacy of an Ultrasound Device in the Management of Acute Acne Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Denise G. Link, PhD, WHNP-BC, CNE, FNAP, Associate Dean, Arizona State University, College of Nursing and Healthcare Innovation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U/S1-SPOT
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ultrasound (Other)
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — ultrasound exposure on acute acne lesions

SUMMARY:
The purpose of this study is to find out how effective and safe an experimental ultrasound device is for treating Acute Acne lesions.

DETAILED DESCRIPTION:
Acne vulgaris is a disease that occurs when oil and dead skin cells clog the pores of the skin. When the skin's pores are clogged, red spots and bumps known as pimples are formed, usually on the face, neck, chest, and back. In adolescents and adults, acne vulgaris is commonly called "acne." Many factors have been associated with acne. One of the factors is the increased production of fatty substances from an enlarged sebaceous gland ("oil gland").

The experimental ultrasonic device uses sound waves (called ultrasonic waves) to heat the acute acne lesion and the surrounding sebaceous ("oil") glands deep in the skin without affecting the surface of the skin. We hope that heating the sebaceous glands will reduce their size and reduce the symptoms of inflamed acne. Using ultrasonic waves to treat acne is investigational.

This is a pilot study. A pilot study is done on a small group of subjects to learn if the device will be effective and safe, before the device is used on a larger group of subjects.

ELIGIBILITY:
Inclusion Criteria:

* female or male subjects,
* greater than 18 years age,
* with acute acne on the face.

Exclusion Criteria:

* pregnancy,
* concomitant skin diseases,
* severe acne,
* antibiotic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Time to clear acute acne lesions | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Denise Link, PhD, Principal Investigator — ASU, College of Nursing and Healthcare Innovation
Locations (1):
- Arizona State University, College of Nursing and Healthcare Innovation, Phoenix, Arizona, United States